CLINICAL TRIAL: NCT02990312
Title: The Effect of Sirolimus Plus Maraviroc on the Expression of Chemokine Receptor 5 (CCR5) and the HIV-1 Viral Reservoir in HIV-Infected Renal Transplant Recipients
Brief Title: Impact of Sirolimus and Maraviroc on CCR5 Expression and the HIV-1 Reservoir in HIV-infected Kidney Transplant Recipients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jennifer Husson, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00072807
Record Dates: First submitted 2016-11-21; First posted 2016-12-13 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Hiv; Kidney Transplant; HIV Reservoir; CCR5
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Sirolimus; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus + Maraviroc (Experimental): Participants will be placed on the combination of Sirolimus and Maraviroc, unless they are already on one of these medications.
  Interventions: Drug: Sirolimus + Maraviroc

INTERVENTIONS:
Drug: Sirolimus + Maraviroc — Patients will be placed on the combination of Sirolimus and Maraviroc starting on Day 0 and followed for 96 weeks during which they will have regular monitoring of both clinical safety labs, Sirolimus levels, and research labs to look at the HIV reservoir, CCR5 density, and immune activation
  Other Names: Rapamycin; Rapamune; Selzentry

SUMMARY:
The purpose of this proof of concept, pilot study is to determine whether the unique combination of the human immunodeficiency virus (HIV) co-receptor antagonist, Maraviroc, and the mammalian target of rapamycin (mTOR) inhibitor, Sirolimus, in HIV-infected kidney transplant recipients has an impact on chemokine receptor 5 (CCR5) density, the HIV-reservoir, or rejection of the transplanted kidney. 15 HIV-infected kidney transplant recipients will be recruited and their immunosuppressant regimen will be changed to include an mTOR inhibitor (such as Sirolimus) unless they are already on one. In addition, Maraviroc will be added to their HIV regimen, unless they are already on Maraviroc. Blood will be taken to measure markers of the HIV reservoir, their CCR5 density and expression, and immune activation.

DETAILED DESCRIPTION:
The study will be a pilot, prospective, single-center, open-label, non-randomized, non-controlled clinical trial. 15 HIV-infected kidney transplant recipients will be enrolled in the study. Recruitment will be conducted through the renal transplant and infectious diseases outpatient clinics at the University of Maryland.

The study will include patients with stable glomerular filtration rates (GFRs) >25 with suppressed HIV with CD4 counts >200. These patients will be recruited from the University of Maryland's transplant nephrology and infectious diseases clinics. The transplant nephrology clinic is a multidisciplinary clinic that incorporates nephrologists, pharmacists to aid in medication management, and coordinators to assist the patients in coordination of care.

All patients will be screened either at the Institute of Human Virology (IHV) Clinical Research Unit or in the transplant nephrology or infectious disease clinics. At this visit, all patients will sign an informed consent as approved by our institutional review board (IRB), have a history and physical examination, and have screening clinical and research labs drawn. Additional requirements will be Trofile testing prior to enrollment. Eligibility will be determined based upon these results.

Study drugs will be prescribed (if the patient is not already taking them) starting on day 0 after an interval history and physical examination is performed and safety labs (and pregnancy tests for women of childbearing potential) are checked. The medications will be filled by the patient's pharmacy, using their insurance as these are both Food and Drug Administration (FDA) approved drugs.

Patients will be initially monitored weekly for sirolimus levels and renal function, until their sirolimus is at the pre-determined (by their transplant nephrologist) steady state. They will then be followed at week 4, and then every 12 weeks while they are on the new medication combination. Safety labs (blood counts, renal and liver function), HIV viral loads, cluster of differentiation 4 (CD4) counts, and rapamycin levels will be reviewed at each of these visits and if not checked within the specified time period these labs will be repeated at the study visit. Patients will also be advised about study adherence and monitored for adverse events.

Safety and adverse event monitoring will occur each study visit. Research nurses will inquire about adverse events that may or may not be related to study drugs. Any unfavorable medical occurrences will be recorded, whether or not considered related to the patient's participation in the research or temporally associated with the patient's participation in the research. Any grade 3 or 4 AEs and all serious adverse events (SAEs) will be reviewed as they occur by the study team. Adverse events (AEs) classified as grade 3 or higher occurring at a frequency greater than that expected by the study team will be reported to the IRB and principal investigator.

The end of treatment visit will occur at week 96. Clinical safety labs (blood counts, renal and liver function), HIV viral load, CD4 counts and rapamycin levels will be performed at this visit if not done in the pre-specified time period. Patients will be given the option, in conjunction with their transplant nephrologist and their infectious disease provider, to discontinue or continue the new medications at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to understand and provide informed consent and comply with the study protocol
2. Diagnosis of HIV infection based on medical record documentation, ELISA and western blot testing, or a record of a detectable HIV viral load
3. Participant is > or = 18 years
4. CD4 T cell count > or = 200 cells per microliter within 16 weeks prior to enrollment
5. Most recent HIV-1 RNA < 50 copies per milliliter within 16 weeks prior to enrollment
6. Participant must be > or = 6 months post-renal transplant
7. GFR >25 for a minimum of 6 months prior to enrollment
8. On a maintenance immunosuppressive regimen for a minimum of 6 months prior to enrollment
9. Female participants of child bearing age must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test within 30 days of enrollment and agree to use contraception during the study

Exclusion Criteria:

1. Proteinuria at screening defined by spot urine protein to creatinine ratio >1000 milligrams per gram
2. The following active opportunistic infections: Ongoing chronic infections such as progressive multifocal leukoencephalopathy (PML), disseminated cryptococcosis, chronic cryptosporidiosis
3. Active malignancy other than superficial skin neoplasms, vulvar intraepithelial neoplasia (VIN), cervical intraepithelial neoplasia (CIN), or anal intraepithelial neoplasia (AIN)
4. Any history of augmented immunosuppression with induction immunosuppression regimens for the treatment of rejection in the 6 months prior to enrollment
5. Known allergy or intolerance to maraviroc or sirolimus
6. Pregnancy or breastfeeding
7. Active substance abuse or mental health concerns that are judged to place a significant limitation on medication adherence by the PI.
8. Triglyceride elevation at screening > 750; or LDL-c > 160 despite medical treatment
9. Use of any investigational drugs within 30 days prior to screening
10. History of serious adverse reactions to macrolide antibiotics, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and abdominal pain.
11. Past or current medical problems not listed above which, at the discretion of the investigator, may pose additional risks from participation in the study, interfere with the participants ability to comply with study requirements or impact the quality or interpretation of data obtained from the study
12. Known contraindication to the use of maraviroc or sirolimus
13. Current and ongoing need for concomitant use of rifampin, rifabutin, rifapentine, St. John's wort, phenytoin, phenobarbital, carbamazepine or dofetilide
14. Any current incompletely healed wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
HIV viral reservoir | 96 weeks
  total cellular HIV DNA

SECONDARY OUTCOMES:
Secondary measures of the HIV viral reservoir | 96 weeks
  Chromosomal HIV DNA
Circulating HIV | 96 weeks
  Ultrasensitive HIV RNA
CCR5 Receptor Density | 96 weeks
  CCR5 receptor density
CCR5 Expression | 96 weeks
  Percentage of T cells expressing CCR5
Acute cellular rejection | 96 weeks
  Incidence of T cell mediated rejection (ACR)
Antibody mediated rejection | 96 weeks
  Incidence of antibody mediated rejection (AMR)
Markers of immune activation/inflammation measured by Ki67 | 96 weeks
  Measurement of Ki67
Markers of immune activation/inflammation measured by cluster of differentiation 38 (CD38) | 96 weeks
  Measurement of CD38
Markers of immune activation/inflammation measured by human leukocyte antigen-antigen D Related (HLA DR) | 96 weeks
  Measurement of HLA DR
Markers of immune activation/inflammation measured by programmed death 1 (PD-1) | 96 weeks
  Measurement of PD-1

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Husson, MD,MPH, Principal Investigator — University of Maryland, College Park
Locations (1):
- Institute of human virology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No